CLINICAL TRIAL: NCT06719518
Title: Performance Evaluation of the ViTrack Continuous Non-invasive Blood Pressure Measurement Device
Status: Not yet recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mehmet Turan, Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-24-0970
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Blood Pressure
Keywords: ViTrack; blood pressure monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- ViTrack device
  Interventions: Device: ViTrack device

INTERVENTIONS:
Device: ViTrack device — In the operating room the ViTrack™ device will be applied the wrist. Monitoring will start in the operating room and will continue throughout the surgery. The device can be worn on either wrist. It will be connected to a power unit that will capture blood pressure data and stream the data to a secure laptop

SUMMARY:
The purpose of this study is to calibrate the ViTrack™ arterial pressure waveform against intra-arterial pressure (IAP) in dynamic clinical settings and to assess the optimized ViTrack™ design to measure and continuously track blood pressure over a wide, clinically-relevant pressure range.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo noncardiac surgery with general or spinal anesthesia
* clinical indication for invasive intra-arterial pressure monitoring
* palpable pulse

Exclusion Criteria:

* difference of greater than 10 mmHg in the left versus right arm oscillometric systolic blood pressure
* Upper extremity arteriovenous hemodialysis shunt
* Upper extremity amputation
* Planned surgical position/draping that precludes access to the wrist
* Wrist distortion or pain from arthritis
* Prior trauma or surgery at the radial artery monitoring site
* Unable to provide informed consent
* Clinical contraindication as determined by the clinical team or study investigators

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: subjects scheduled to undergo noncardiac surgery with likely invasive arterial pressure monitoring will be included will be included
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Comparison of Diastolic Blood Pressure | From start of surgery up to 24 hours after surgery
  255 time points compared across continuous blood pressure (mmHg)
Comparison of Systolic Blood Pressure | From start of surgery up to 24 hours after surgery
  255 time points compared across continuous blood pressure (mmHg)

SECONDARY OUTCOMES:
Number of participants who show signs of Skin Irritation | From start of surgery up to 72 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Turan, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No